CLINICAL TRIAL: NCT05387226
Title: A Sing-Arm, Open Clinical Pharmacology Study of Intravenous Injection of Oncolytic Virus Injection (RT-01) in Patients With Relapsed or Refractory T-cell Lymphoma
Brief Title: Intravenous Injection of Oncolytic Virus Injection (RT-01) in Patients With Relapsed or Refractory T-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Zhang Feng, MD, Deputy Director of Hematology, The First Affiliated Hospital of Bengbu Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LWY21076CBY3
Record Dates: First submitted 2022-05-07; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: T-cell Lymphoma; Virus; Intravenous Injection
MeSH Terms: conditions — Lymphoma, T-Cell; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncolytic Virus Injection(RT-01) (Experimental): RT-01 will be administered intravenously
  Interventions: Biological: Oncolytic Virus Injection(RT-01)

INTERVENTIONS:
Biological: Oncolytic Virus Injection(RT-01) — RT-01 will be administered intravenously on day 1 and 6, and every 8 weeks thereafter (up to 6 times)

SUMMARY:
This is a single-arm, open-label, clinical pharmacology study to evaluate safety and efficacy of oncolytic virus injection(RT-01) in patients with Relapsed or Refractory T-cell Lymphoma. The purpose of this study is to evaluate the safety and tolerability, antitumor activity, The immunoreactivity, The immunogenicity, pharmacokinetics and virus shedding of RT-01.

DETAILED DESCRIPTION:
This is an investigator initiated , single-arm, open-label clinical pharmacology study of RT-01 given via Intravenous injection in patients with advanced solid tumors. RT-01 will be administered on days 1 and 6, and every 8 weeks thereafter (up to 6 times).

This study is planned to enroll 6 patients with Relapsed or Refractory T-cell Lymphoma.

The purpose of this study is to assess the safety and tolerability, antitumor activity, The immunoreactivity, The immunogenicity, pharmacokinetics and virus shedding of RT-01.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years.
2. The following of typesRelapsed T-cell lymphoma (TCL): peripheral T-cell lymphoma (PTCL) [peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell (ALCL)], and cutaneous TCL (CTCL) of mycosis fungoides (MF).
3. Patients have received at least 1-line systemic treatment in the past and who have relapsed or are refractory: failed to achieve complete remission (CR) or disease progression (PD) after CR, ineligible for autologous hematopoietic stem cell transplantation (ASCT) or PD after ASCT.
4. There is at least one measurable lesion without previous local treatment, which the long axis of the intranodal lesion is >15 mm or extranodal lesion >10 mm According to Lugano 2014 criteria.
5. Patients Eastern Cooperative Oncology Group (ECOG) physical status score must be 0 or 1.
6. Life expectancy≥3 months et al.

Exclusion Criteria:

1. Subjects with brain metastasis and/or clinically history tumor brain of metastasis;
2. Subjects who have received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc within 2 weeks before RT-01 administration;
3. Subjects who have participate in another interventional study within 4 weeks before RT-01 administration;
4. Subjects who have had major surgery within 4 weeks before RT-01 administration.
5. Patients in any condition requiring systemic treatment with corticosteroids (prednisone > 10 mg/day or equivalent of the similar drug) or other immunosuppressive agents within 14 days before RT-01 administration, but currently or previously treated with any of the following steroid regimens, were included: Topical, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption; Prophylactic short-term use of corticosteroids;
6. Subjects who have participate in another oncolytic virus study within 8 weeks before RT-01 administration;
7. Subjects received live vaccines within 7 days before RT-01 administration;
8. Subjects received Antiviral drugs within 2 weeks, long-acting interferon within 4 weeks before RT-01 administration# 9.Subjects with adverse reactions caused by previous anti-tumor treatment not recovered to (CTCAE 5.0) grade 1 (except alopecia);

10.Subjects who have uncontrolled active infection; 11.Subjects with known positive history of human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS); 12.Subjects who have active hepatitis; 13.Subjects who have serious cardiovascular system disorders history; 14.Clinically uncontrollable third space effusion,are considered unsuitable for this study in the opinion of the investigator; 15.Subjects with active autoimmune diseases or history of autoimmune diseases that may relapse; et al.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Graded according to the NCI CTCAE version 5.0.
To evaluate objective Response Rate (ORR) of the antitumor activity | Up to 2 years
  To assessed per Lugano and Lyric
To evaluate the disease control rate (DCR) of the antitumor activity | Up to 2 years
  To assessed per Lugano and Lyric
The changes of the immunoreactivity during treatment | Up to 28 days
  Peripheral blood T lymphocyte subtype
To evaluate the immunogenicity of RT-01 | Up to 28 days
  Antiviral antibody
To evaluate the viral shedding of RT-01 | 8 weeks after last dose
  Viral RNA
The Cmax of Viral RNA | 8 weeks after last dose
  The maximum RNA peak concentration
The Tmax of Viral RNA | 8 weeks after last dose
  The time of maximum RNA peak concentration

IPD SHARING:
Plan to Share IPD: No